CLINICAL TRIAL: NCT02968108
Title: A Randomized Double-blind Pharmacokinetic Study of Ustekinumab in Pediatric Subjects With Moderately to Severely Active Crohn's Disease
Brief Title: A Pharmacokinetic Study of Ustekinumab in Pediatric Subjects With Moderately to Severely Active Crohn's Disease
Acronym: STELARA
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR108233; CNTO1275CRD1001 (Other: Janssen Research & Development, LLC); 2016-001956-22 (EudraCT Number)
Record Dates: First submitted 2016-10-24; First posted 2016-11-18 (Estimated); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Crohn Disease
MeSH Terms: conditions — Crohn Disease | interventions — Ustekinumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group1: Ustekinumab Dose Regimen 1 (Experimental): Subjects will receive a single intravenous (IV) induction dose of 3 milligram per kilogram (mg/kg) for subjects less than < 40 kilogram (kg) or 130 milligram (mg) for subjects greater than or equal to >= 40 kg at Week 0 followed by subcutaneous (SC) maintenance dose of 2 mg/kg for subjects < 40 kg or 90 mg for subjects >= 40 kg at week 8.
  Interventions: Drug: Ustekinumab
- Group2: Ustekinumab Dose Regimen 2 (Experimental): Subjects will receive a single Intravenous (IV) dose of 9 mg/kg for subjects <40 kg or 390 mg for subjects >= 40 kg at Week 0 followed by SC maintenance dose of 2 mg/kg for subjects <40 kg or 90 mg for subjects >= 40 kg at week 8.
  Interventions: Drug: Ustekinumab

INTERVENTIONS:
Drug: Ustekinumab — Subjects will receive a single IV administration of ustekinumab (3 mg/kg for subjects <40 kg or 130 mg for subjects >= 40 kg in Group 1 and 9 mg/kg for subjects < 40 kg or 390 mg for subjects >= 40 kg in group 2) at week 0 followed by SC administration of ustekinumab (2 mg/kg for subjects < 40 kg or 90 mg for subjects >= 40 kg at Week 8.

SUMMARY:
The purpose of this study is to evaluate the pharmacokinetics (PK) of ustekinumab in subjects from 2 through less than (<) 18 years old in the USA, or 6 through less than (<) 18 years old in other countries and determine if it is similar to that observed in adults with moderately to severely active Crohn's disease (CD). Also to assess the safety, immunogenicity and efficacy of ustekinumab in the treatment of moderately to severely active CD. The main part of the study continues to Week 16, at which point all subjects who are receiving benefit from ustekinumab maintenance therapy (as determined by the investigator) are eligible to enter the long-term extension (LTE) and continue to receive ustekinumab. The study extension ends at Week 268 or upon availability of the LTE basket study (CNTO1275ISD3001) whichever occurs first. If participants do not consent/assent to the LTE basket study, they will continue safety follow-up for approximately 20 weeks after the last study agent administration.

ELIGIBILITY:
Inclusion Criteria:

* Be a pediatric subject 2 to less than (<) 18 years old in the US, 6 to <18 years old elsewhere, of either gender with a body weight of greater than or equal to (>=) 10 kilogram (kg)
* Have Crohn's disease (CD) or fistulizing CD of at least 3 months duration, with active colitis, ileitis, or ileocolitis, confirmed at any time in the past by radiography, histology, and/or endoscopy
* Must have moderately to severely active CD defined by: Baseline pediatric Crohn's disease activity index (PCDAI) score of greater than (>)30 and at least one of the following: An abnormal C-reactive protein (CRP) >0.3 milligram per deciliter (mg/dL) or 3.0 milligram per liter (mg/L) at screening) or fecal calprotectin >250 milligram per kilogram (mg/kg) at screening or ileocolonoscopy with evidence of active CD (defined as ulcerations in the ileum and/or colon) during screening into this study including at the baseline visit
* Prior or current medication for CD must include at least 1 of the following: Current treatment with at least 1 of the following therapies: oral corticosteroids, the immunomodulators azathioprine, 6-MP, or methotrexate, or currently have or have had a history of corticosteroid dependency, or have a history of failure to respond to, or tolerate, at least 1 of the following therapies including oral or IV corticosteroids or the immunomodulators 6-mercaptopurine, azathioprine, or methotrexate,or have required more than 3 courses of oral or IV corticosteroids in the past year
* Have negative stool results for enteric pathogens. Stool studies must include a stool culture and Clostridium difficile toxin assay. These must have been performed during screening or the current episode of disease exacerbation as long as the stool studies were performed within 4 months prior to the first administration of study agent

Exclusion Criteria:

* Has complications of CD such as symptomatic strictures or stenosis, short gut syndrome, or any other manifestation that might be anticipated to require surgery, could preclude the use of the PCDAI to assess response to therapy, or would possibly confound the ability to assess the effect of treatment with ustekinumab
* Currently has or is suspected to have an abscess. Recent cutaneous and perianal abscesses are not exclusionary if drained and adequately treated at least 3 weeks prior to baseline, or 8 weeks prior to baseline for intra-abdominal abscesses, provided that there is no anticipated need for any further surgery. Participant with active fistulas may be included if there is no anticipation of a need for surgery and there are currently no abscesses identified
* Has had any kind of bowel resection within 6 months or any other intra-abdominal surgery within 3 months prior to baseline
* Has a draining (that is (i.e.), functioning) stoma or ostomy
* Presence or history of any malignancy including presence or history of lymphoproliferative disease including lymphoma, or signs and symptoms suggestive of possible lymphoproliferative disease, such as lymphadenopathy of unusual size or location (example, nodes in the posterior triangle of the neck, infraclavicular, epitrochlear, or periaortic areas), or clinically significant hepatomegaly or splenomegaly

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 45 (Actual)
Dates: Start 2017-01-18 (Actual); Primary Completion 2018-09-19 (Actual); Study Completion 2022-03-18 (Actual)

PRIMARY OUTCOMES:
Serum Ustekinumab Concentrations Over Time | Up to Week 16
  Serum samples will be collected to measure seum concentrations of Ustekinumab.

SECONDARY OUTCOMES:
Clinical Response as Measured by the Pediatric Crohn's Disease Activity Index (PCDAI) Score | Week 6
  Clinical Response is defined as greater than or equal to (>=) 15-point reduction from baseline in the total Pediatric Crohn's Disease Activity Index (PCDAI) score, accompanied by a total PDCAI score of less than or equal to (<=) 30 points. PCDAI is an index used to measure disease activity of pediatric patients with Crohn's Disease assessing abdominal pain, stool frequency, patient functioning, hematocrit, erythrocyte sedimentation rate, albumin, weight, height, abdominal tenderness or mass, perirectal disease, and extraintestinal manifestations. It ranges from 0 to 100; higher scores indicate more active disease.
Clinical Remission as Measured by the Pediatric Crohn's Disease Activity Index (PCDAI) Score | Week 8
  Clinical remission is defined as PCDAI score of less than or equal to (<=) 10. PCDAI is an index used to measure disease activity of pediatric patients with Crohn's Disease assessing abdominal pain, stool frequency, patient functioning, hematocrit, erythrocyte, sedimentation rate, albumin, weight, height, abdominal tenderness or mass, perirectal disease, and extraintestinal manifestations. It ranges from 0 to 100; higher scores indicate more active disease.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (26):
- United States (9):
  - Cedars Sinai Medical Center, Los Angeles, California
  - Connecticut Childrens Medical Center, Hartford, Connecticut
  - Emory University, Atlanta, Georgia
  - Children's Center For Digestive Healthcare, Llc, Atlanta, Georgia
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - Mayo Clinic, Rochester, Minnesota
  - Mount Sinai, New York, New York
  - Childrens Hospital Of Philadelphia, Philadelphia, Pennsylvania
  - Center For Digestive Health Systems-Greenville, Greenville, South Carolina
- Belgium (5):
  - Universitair Kinderziekenhuis Koningin Fabiola, Brussels
  - Cliniques Universitaires Saint Luc, Brussels
  - UZ Gent, Ghent
  - UZ Brussel, Jette
  - UZ Leuven, Leuven
- Canada (5):
  - Stollery Children's Hospital, Edmonton, Alberta
  - British Columbia Children's Hospital, Vancouver, British Columbia
  - Children's Hospital of Western Ontario, London, Ontario
  - Hospital For Sick Children, Toronto, Ontario
  - Centre Hospitalier Sainte Justine, Montreal, Quebec
- France (2):
  - Hôpital Necker, Paris
  - Hôpital Robert Debré, Paris
- Germany (2):
  - Dr. von Haunersches Kinderspital, Munich
  - HELIOS Klinikum Wuppertal GmbH, Wuppertal
- Poland (3):
  - Instytut Centrum Zdrowia Matki Polki, Lodz
  - WIP Warsaw IBD Point Profesor Kierkus, Warsaw
  - Uniwersytecki Szpital Kliniczny im Jana Mikulicza Radeckiego we Wroclawiu, Wroclaw

REFERENCES:
- [Derived] Hasskamp J, Meinhardt C, Timmer A. Anti-IL-12/23p40 antibodies for induction of remission in Crohn's disease. Cochrane Database Syst Rev. 2025 May 13;5(5):CD007572. doi: 10.1002/14651858.CD007572.pub4. PMID 40357993